CLINICAL TRIAL: NCT03310359
Title: A Double-blinded, Placebo-controlled, Clinical Trial of Insulin-sensitizing, Anti-inflammatory and Anti-oxidant Activities of Astaxanthin in Insulin-resistant Subjects
Brief Title: Clinical Trial of Anti-oxidant Astaxanthin in Insulin-resistant Subjects
Acronym: Astaxanthin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 151542
Record Dates: First submitted 2016-11-02; First posted 2017-10-16 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: A double-blinded, placebo controlled, Clinical Trial of Insulin-Sensitizing, Anti-Inflammatory and Anti-oxidant activities of Astaxanthin in Insulin-resistant Subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astaxanthin (12 mg) (Active Comparator): Subjects will be given capsules containing a set oral dose of astaxanthin (12 mg) and instructed to take two capsules each morning after (up to 1 hr) the morning meal for a total of up to 24 weeks (168 days on study drug).
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): Subjects will be given capsules containing placebo and instructed to take two capsules each morning after (up to 1 hr) the morning meal for a total of up to 24 weeks (168 days on study drug).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin — The agent to be tested is astaxanthin, isolated from H. pluvialis following GMP standards. A GRAS notice (GRN000294) was accepted by the Food and Drug Administration (FDA) in January 2010. Agent is stored in capsules at room temperature.
  Other Names: Haematococcus pluvialis
  Arms: Astaxanthin (12 mg)
Other: Placebo — Matching placebo pill
  Arms: Placebo

SUMMARY:
Astaxanthin is a natural compound, present in many foodstuffs and available as a nutritional supplement that has been shown to have beneficial effects on many of the features of insulin resistance/glucose intolerance, at least in animals. The goal of this project is to provide a validation of astaxanthin effects on metabolic regulation in humans and their mechanism(s) of action, to determine if astaxanthin could have any value as a "neutraceutical" to help improve regulation of glucose and fat metabolism in subjects with insulin resistance/ glucose intolerance.

DETAILED DESCRIPTION:
Astaxanthin is a molecule of the carotenoid class that is abundant in marine animals and plants, with the algae Haematococcus pluvialis being a particularly rich source. Astaxanthin is a potent anti-oxidant with a unique property of being able to insert into membranes and lipid bilayers. Astaxanthin has also been shown to be a potent anti-inflammatory agent. As oxidative stress and inflammation are present in individuals with insulin resistance, astaxanthin offers promise as a potential therapeutic for this patient population.

There are a number of formulations of astaxanthin that are available for use in humans. With regard to controlled studies in humans, astaxanthin has been given at doses as high as 40 mg/day for periods from 2 to 12 weeks. Improvements in inflammation and oxidative stress were frequently observed. With regard to metabolic regulation, improvements have been seen in HDL and LDL levels, while others have found no changes. Glucose and insulin levels appear to be unaltered: This lack of effect may be due to only healthy, though in some cases overweight or obese, subjects being studied. In none of these studies, were any abnormal safety lab values or adverse events reported. One of the intents of the current project is to perform more detailed metabolic characterization of astaxanthin treatment effects in research participants with insulin resistance/glucose intolerance.

The hyperinsulinemic-euglycemic glucose clamp procedure (HEC) will be used to assess insulin sensitivity and responsiveness by measuring glucose disposal rate (GDR). Investigators will also perform Oral Glucose Tolerance Tests (OGTT), indirect calorimetry (IDC), and 24 hour measurement of ambulatory blood pressure (ABPM).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years (inclusive)
* Both males and females
* If female, must be post-menopausal or not capable of becoming pregnant
* Able to give informed consent to the procedures
* Dyslipidemia - [TG]>150, or [LDL]>100 or [HDL]<40 for males, <50 for females or taking a statin or fibrate
* BMI = 25-39
* Impaired fasting glucose 95>[FG]<125 and/or elevated HbA1c (5.7-6.4%)
* Concomitant medication use stable for 30 days prior to screening visit (Acceptable medications: anti-hypertensive if blood pressure criteria met statins or fibrates)

Exclusion Criteria:

* Type 2 diabetes
* Type 1 diabetes
* Pregnant
* Younger than 18 or older than 75 years of age.
* Clinically significant abnormalities in liver (> 3x ULN) or kidney function (eGFR < 30)
* Myocardial Infarction (MI) (within 6 months of screening)
* Stroke (within 6 months of screening)
* Blood pressure (BP) >160 mmHg Systolic and >100 mmHg Diastolic
* The following medications are exclusionary: thiazolidinediones, any steroids, anti-depressants, weight loss, and OTC antioxidants (if taking OTC antioxidant supplements, subjects must be willing to stop taking them immediately upon site verifying that the subject qualifies for enrollment and for the duration of the entire study. Some OTC antioxidants may be acceptable upon approval by the Principal Investigator.)
* Other disease, besides type 2 diabetes, influencing carbohydrate metabolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | 6 months
  Change from baseline insulin sensitivity during hyperinsulinemic/euglycemic clamp at 6 months.

SECONDARY OUTCOMES:
Change in lipid control | 6 months
  Change from baseline suppression of Free Fatty Acids (FFAs) during hyperinsulinemic/euglycemic clamp at 6 months.
Change in fasting glucose | 6 months
  Change from baseline fasting glucose at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Pettus, MD, Principal Investigator — UCSD
Locations (1):
- Altman Clinical and Translational Research Institute (ACTRI), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No